CLINICAL TRIAL: NCT04224688
Title: A Phase 3 Multicenter, Double-Blind, Randomized, Placebo-Controlled Study to Evaluate the Efficacy, Safety, and Tolerability of Rozanolixizumab in Adult Study Participants With Persistent or Chronic Primary Immune Thrombocytopenia (ITP)
Brief Title: A Study to Assess the Efficacy, Safety, and Tolerability of Rozanolixizumab in Adult Study Participants With Persistent or Chronic Primary Immune Thrombocytopenia (ITP)
Acronym: myOpportunITy2
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Strategic Business Decision; Not a safety decision
Sponsor: UCB Biopharma SRL (Industry)
Responsible Party: Sponsor
Organization: UCB Pharma (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TP0006; 2019-003451-11 (EudraCT Number)
Record Dates: First submitted 2020-01-08; First posted 2020-01-13 (Actual); Results first posted 2023-08-08 (Actual); Last update posted 2023-08-08 (Actual); Status verified 2023-08

CONDITIONS: Primary Immune Thrombocytopenia
Keywords: ITP; UCB7665; Rozanolixizumab; Primary Immune Thrombocytopenia
MeSH Terms: conditions — Purpura, Thrombocytopenic, Idiopathic | interventions — rozanolixizumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Investigators are blinded to the treatment code, they will see the platelet values.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Rozanolixizumab (Experimental): Study participants randomized to this arm will receive fixed-unit doses of rozanolixizumab across body weight tiers at pre-specified time points during the Treatment Period. Doses will be adjusted based on platelet count values or medical needs.
  Interventions: Drug: Rozanolixizumab
- Placebo (Placebo Comparator): Study participants randomized to this arm receive placebo at pre-specified time points during the Treatment Period.
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Rozanolixizumab — Study participants receive rozanolixizumab by subcutaneous infusion at pre-specified time points.
  Other Names: UCB7665
  Arms: Rozanolixizumab
Other: Placebo — Study participants receive placebo by subcutaneous infusion at pre-specified time points.
  Arms: Placebo

SUMMARY:
The purpose of this study is to demonstrate the clinical efficacy of rozanolixizumab in maintenance treatment and assess safety and tolerability of rozanolixizumab in adult study participants with primary immune thrombocytopenia (ITP).

ELIGIBILITY:
Inclusion Criteria:

* Study participant must be ≥18 years of age at the time of the Screening Visit
* Study participant has a diagnosis of persistent (>3 months duration) or chronic (>12 months duration) primary immune thrombocytopenia (ITP) at the Screening Visit
* Study participant has a documented intolerance or insufficient response to two or more appropriate standard of care ITP treatments prior to Screening
* Study participants must have prior history of a response to a previous ITP therapy.
* If taking allowed drugs, study participant must be on stable doses during defined time periods prior to Baseline (Day 1)
* Study participant has a documented history of low platelet count (<30×10^9/L) prior to Screening
* Study participant has a platelet count measurement at Screening and at Baseline (Day 1) with an average of the two <30×10^9/L and no single count may be >35×10^9/L (using local laboratories)
* Study participant has a current or history of a peripheral blood smear consistent with ITP
* Study participants may be male or female:

  1. A male participant must agree to use contraception during the Treatment Period and for at least 3 months after the final dose of study treatment and refrain from donating sperm during this period
  2. A female participant is eligible to participate if she is not pregnant as confirmed by a negative serum pregnancy test and not planning to get pregnant during the participation in the study, not breastfeeding, and at least one of the following conditions applies:

Not a woman of childbearing potential (WOCBP) OR A WOCBP who agrees to follow the contraceptive guidance during the Treatment Period and for at least 3 months after the dose of study treatment

Exclusion Criteria:

* Participant has a history of arterial or venous thromboembolism (eg, stroke, transient ischemic attack, myocardial infarction, deep vein thrombosis or pulmonary embolism) within the 6 months prior to randomization or requires current anticoagulant treatment
* Study participant has clinically significant bleeding that warrants immediate platelet adjustment (eg, menorrhagia with significant drop in hemoglobin)
* Study participant has a known hypersensitivity to any components of the study medication or any other anti-neonatal Fc receptor (FcRn) medications
* Study participant has evidence of a secondary cause of immune thrombocytopenia (clear association with other medical conditions eg, of untreated H. pylori infection, leukemia, lymphoma, common variable immunodeficiency, systemic lupus erythematosus, autoimmune thyroid disease or is drug induced), participant has a multiple immune cytopenia (eg, Evan's syndrome) etc.
* Study participant has a clinically relevant active infection (eg, sepsis, pneumonia, or abscess) in the opinion of the investigator, or had a serious infection (resulting in hospitalization or requiring parenteral antibiotic treatment) within 6 weeks prior to the first dose of investigational medicinal product (IMP)
* Study participant with a known tuberculosis (TB) infection, at high risk of acquiring TB infection, or latent tuberculosis infection (LTBI), or current/history of nontuberculous mycobacterial infection (NTMBI)
* Study participant has a history of a major organ transplant or hematopoietic stem cell/marrow transplant
* Study participant has experienced intracranial bleed in the last 6 months prior to the Screening Visit
* Study participant has a history of coagulopathy disorders other than ITP
* Study participant with current or medical history of immunoglobulin A (IgA) deficiency, or a measurement of IgA <50 mg/dL at the Screening Visit
* Study participant has undergone a splenectomy in the 2 years prior to the Baseline Visit

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2020-06-03 (Actual); Primary Completion 2022-04-25 (Actual); Study Completion 2022-05-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: UCB Cares, Study Director — 001 844 599 2273
Locations (29):
- United States (2):
  - Tp0006 50412, St. Petersburg, Florida
  - Tp0006 50243, Boston, Massachusetts
- Bulgaria (2):
  - Tp0006 40189, Plovdiv
  - Tp0006 40008, Sofia
- China (9):
  - Tp0006 20201, Bengbu
  - Tp0006 20189, Changchun
  - Tp0006 20188, Changsha
  - Tp0006 20186, Changzhou
  - Tp0006 20179, Fuzhou
  - Tp0006 20187, Hangzhou
  - Tp0006 20177, Jinan
  - Tp0006 20185, Jinan
  - Tp0006 20194, Wuxi
- Tp0006 40364, Lille, France
- Germany (2):
  - Tp0006 40369, Berlin
  - Tp0006 40366, Rostock
- Poland (2):
  - Tp0006 40219, Słupsk
  - Tp0006 40223, Warsaw
- Russia (3):
  - Tp0006 20052, Moscow
  - Tp0006 20054, Moscow
  - Tp0006 20053, Saint Petersburg
- Spain (3):
  - Tp0006 40231, Madrid
  - Tp0006 40268, Madrid
  - Tp0006 40381, Zaragoza
- Taiwan (2):
  - Tp0006 20094, Tainan
  - Tp0006 20095, Taipei
- Ukraine (2):
  - Tp0006 20061, Cherkasy
  - Tp0006 20064, Kyiv
- Tp0006 40239, Leeds, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Data from this trial may be requested by qualified researchers six months after product approval in the US and/or Europe, or global development is discontinued, and 18 months after trial completion. Investigators may request access to anonymized individual patient-level data and redacted trial documents which may include: analysis-ready datasets, study protocol, annotated case report form, statistical analysis plan, dataset specifications, and clinical study report. Prior to use of the data, proposals need to be approved by an independent review panel at www.Vivli.org and a signed data sharing agreement will need to be executed. All documents are available in English only, for a prespecified time, typically 12 months, on a password protected portal. This plan may change if the risk of re-identifying trial participants is determined to be too high after the trial is completed; in this case and to protect participants, individual patient-level data would not be made available.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Data from this study may be requested by qualified researchers six months after product approval in the US and/or Europe or global development is discontinued, and 18 months after trial completion.
Access Criteria: Qualified researchers may request access to anonymized IPD and redacted study documents which may include: raw datasets, analysis-ready datasets, study protocol, blank case report form, annotated case report form, statistical analysis plan, dataset specifications, and clinical study report. Prior to use of the data, proposals need to be approved by an independent review panel at www.Vivli.org and a signed data sharing agreement will need to be executed. All documents are available in English only, for a pre-specified time, typically 12 months, on a password protected portal.
URL: https://www.Vivli.org

REFERENCES:
- See also: FDA Safety Alerts and Recalls — http://www.fda.gov/Safety/MedWatch/SafetyInformation/default.htm

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study started to enroll study participants in June 2020 and terminated in May 2022.
Pre-assignment Details: Participant Flow refers to the Randomized Set.
Groups:
- Placebo: Participants received a fixed-unit starting dose of placebo subcutaneous (sc) infusion matched to rozanolixizumab Dose A on Day 1. Following the initial dose, participants received a fixed-unit dose of placebo sc infusion matched to rozanolixizumab Dose B every 2 weeks until Week 23. Participants were followed up to a maximum of Week 31.
- Rozanolixizumab: Participants received a fixed-unit starting dose of rozanolixizumab sc infusion equivalent to Dose A on Day 1. Following the initial dose, participants received a fixed-unit dose of rozanolixizumab sc infusion equivalent to Dose B every 2 weeks until Week 23. After protocol amendment 3, the starting dose was removed and the frequency of administration of the Dose B was changed to weekly. Participants were followed up to a maximum of Week 31.
Period: Overall Study
Arm/Group | Placebo | Rozanolixizumab
Started | 10 | 20
Completed | 8 | 13
Not Completed | 2 | 7
Not completed — Withdrawal by Subject | 1 | 3
Not completed — Lack of Efficacy | 1 | 1
Not completed — Adverse event, not fatal | 0 | 2
Not completed — COVID-19 | 0 | 1

BASELINE CHARACTERISTICS:
Population: Baseline Characteristics refer to Randomized Set which consisted of all enrolled study participants who were randomized.
Groups:
- Placebo: Participants received a fixed-unit starting dose of placebo sc infusion matched to rozanolixizumab Dose A on Day 1. Following the initial dose, participants received a fixed-unit dose of placebo sc infusion matched to rozanolixizumab Dose B every 2 weeks until Week 23. Participants were followed up to a maximum of Week 31.
- Total: Total of all reporting groups
Arm/Group | Placebo | Rozanolixizumab | Total
Number analyzed (Participants) | 10 | 20 | 30
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 1 | 1
  Between 18 and 65 years | 10 | 17 | 27
  >=65 years | 0 | 2 | 2
Age, Continuous [Mean (Standard Deviation); unit: years] | 41.9 (14.5) | 42.3 (15.7) | 42.2 (15.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 13 | 19
  Male | 4 | 7 | 11
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 3 | 6 | 9
  White | 7 | 13 | 20
  Missing | 0 | 1 | 1
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 2 | 2
  Not Hispanic or Latino | 10 | 18 | 28
  Missing | 0 | 0 | 0
Platelet count [Mean (Standard Deviation); unit: cells*10^9/L] | 14.10 (7.77) | 14.65 (8.18) | 14.46 (7.91)

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Durable Clinically Meaningful Platelet Response of ≥50×10^9/L, for at Least 8 Out of 12 Weeks During the Last 12 Weeks
Description: Percentage of Participants With Durable Clinically Meaningful Platelet Response of ≥50×10^9/L, for at least 8 out of 12 weeks during the last 12 weeks were reported.
Time Frame: During the last 12 weeks (Week 13 to Week 25)
Population: Randomized Set consisted of all enrolled study participants who were randomized. No formal analysis was carried out as the program was terminated.
Measure: Number; unit: Percentage of participants
Arm/Group | Placebo | Rozanolixizumab
Number analyzed (Participants) | 10 | 20
Percentage of participants | 0 | 5.0

2. Secondary Outcome: Cumulative Number of Weeks With Clinically Meaningful Platelet Response of ≥50×10^9/L Over the 24-week Treatment Period
Description: Total number of weeks with platelet counts ≥50×10^9/L over the 24-week Treatment Period of the study (Week 1 to Week 25) were reported.
Time Frame: Week 1 up to Week 25
Population: Randomized Set consisted of all enrolled study participants who were randomized.
Measure: Median (Full Range); unit: Weeks
Arm/Group | Placebo | Rozanolixizumab
Number analyzed (Participants) | 10 | 20
Weeks | 0.0 [0 to 10] | 1.0 [0 to 18]

3. Secondary Outcome: Time to First Clinically Meaningful Platelet Response (CMPR) of ≥50×10^9/L: Time From Starting Treatment to Achievement of First Response of ≥50×10^9/L
Description: Time from starting treatment to achievement of first Clinically Meaningful Platelet Response of ≥50×10^9/L was defined as date of first clinically meaningful response - date of first treatment + 1. Median was calculated based upon the Kaplan-Meier estimate.
Time Frame: Time from starting treatment to achievement of first response of ≥50×10^9/L (up to Week 25)
Population: Randomized Set consisted of all enrolled study participants who were randomized.
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | Placebo | Rozanolixizumab
Number analyzed (Participants) | 10 | 20
Days | NA [4.0 to NA] — NA for median signifies that the probability of participants achieving a CMPR did not reach 0.5 so the Kaplan-Meier median could not be estimated. NA signifies that upper confidence limit for placebo is not provided for the 95% CI of the median time to first CMPR as there is no time at which the upper bound of the CI for the Kaplan-Meier estimator is less than or equal to 0.5. | 8.0 [5.0 to NA] — NA signifies that upper confidence limit for rozanolixizumab is not provided for the 95% CI of the median time to first CMPR as there is no time at which the upper bound of the CI for the Kaplan-Meier estimator is less than or equal to 0.5.

4. Secondary Outcome: Percentage of Participants With Clinically Meaningful Platelet Response of ≥50×10^9/L by Day 8
Description: Clinically meaningful platelet response was defined as platelet count of ≥50×10^9/L.
Time Frame: Baseline to Day 8
Population: Randomized Set consisted of all enrolled study participants who were randomized.
Measure: Number; unit: Percentage of participants
Arm/Group | Placebo | Rozanolixizumab
Number analyzed (Participants) | 10 | 20
Percentage of participants | 10.0 | 45.0

5. Secondary Outcome: Percentage of Participants With Response Defined as Platelet Count ≥30*10^9/L and at Least Doubling of Baseline, at Least 2 Separate Occasions at Two Adjacent Nominal Visits at Least 7 Days Apart, and Absence of Bleeding
Description: Response was defined as platelet count ≥30*10^9/L and at least doubling of baseline, at least 2 separate occasions at two adjacent nominal visits at least 7 days apart, and absence of bleeding.
Time Frame: From Baseline during Treatment Period (up to Week 25)
Population: Randomized Set consisted of all enrolled study participants who were randomized.
Measure: Number; unit: Percentage of participants
Arm/Group | Placebo | Rozanolixizumab
Number analyzed (Participants) | 10 | 20
Percentage of participants | 10.0 | 20.0

6. Secondary Outcome: Time to First Rescue Therapy
Description: Time to first rescue therapy was defined as date of first rescue therapy use - date of first treatment + 1. Median was calculated based upon the Kaplan-Meier estimate.
Time Frame: From Baseline to first rescue therapy (up to Week 25)
Population: Randomized Set consisted of all enrolled study participants who were randomized.
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | Placebo | Rozanolixizumab
Number analyzed (Participants) | 10 | 20
Days | NA [4.0 to NA] — NA for median signifies that the probability of participants requiring rescue medication did not reach 0.5 so the Kaplan-Meier median could not be estimated. NA signifies that upper confidence limit for placebo is not provided for the 95% CI of the median time to rescue therapy as there is no time at which the upper bound of the CI for the Kaplan-Meier estimator is less than or equal to 0.5. | NA [46.0 to NA] — NA for median signifies that the probability of participants requiring rescue medication did not reach 0.5 so the Kaplan-Meier median could not be estimated. NA signifies that upper confidence limit for rozanolixizumab is not provided for the 95% CI of the median time to rescue therapy as there is no time at which the upper bound of the CI for the Kaplan-Meier estimator is less than or equal to 0.5.

7. Secondary Outcome: Change From Baseline to Week 25 in Primary Immune Thrombocytopenia Patient Assessment Questionnaire (ITP-PAQ) Symptoms Score
Description: The ITP-PAQ Version 1 is a 44 item disease-specific Health-Related Quality of Life questionnaire developed for use in adults with chronic ITP. It includes 10 scales, Four of the scales measure physical health: Symptoms (6 items), Bother (3 items), Fatigue (4 items), and Activity (2 items). Two of the scales measure emotional health: Fear (5 items) and Psychological (5 items) Health. The remaining four scales measure other aspects of quality of life (QOL): Work QOL (4 items), Social QOL (4 items), Women's Reproductive QOL (6 items) and Overall QOL (5 items). Each item is rated on a Likert-type scale containing 4 to 7 responses. All item scores are transformed to a 0 to 100 continuum and are weighted equally to derive individual scale scores and the total score (0-100) is calculated as per the formula: Sum of item scores within the scale/raw sum range*100. Higher scores indicate better health status.
Time Frame: From Baseline during Treatment Period (up to Week 25)
Population: Randomized Set consisted of all enrolled study participants who were randomized. Here, Number of Participants analyzed signifies those participants who were evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Rozanolixizumab
Number analyzed (Participants) | 8 | 12
units on a scale | -0.5 (17.0) | 4.2 (12.9)

8. Secondary Outcome: Percentage of Participants With Treatment-emergent Adverse Events (TEAEs)
Description: An adverse event (AE) is any untoward medical occurrence in a patient or clinical study participant, temporally associated with the use of investigational medicinal product (IMP), whether or not considered related to the IMP. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease (new or exacerbated) temporally associated with the use of IMP. TEAEs are defined as AEs starting after the time of first IMP administration up to and including 8 weeks (56 days) after the final dose.
Time Frame: From Baseline to end of Safety Follow-Up Period (up to Week 31)
Population: Safety set included all randomized study participants who received at least one dose of IMP.
Measure: Number; unit: Percentage of participants
Arm/Group | Placebo | Rozanolixizumab
Number analyzed (Participants) | 10 | 20
Percentage of participants | 60.0 | 95.0

9. Secondary Outcome: Percentage of Participants With TEAEs Leading to Withdrawal of Investigational Medicinal Product (ie, Study Discontinuation)
Description: An AE is any untoward medical occurrence in a patient or clinical study participant, temporally associated with the use of IMP, whether or not considered related to the IMP. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease (new or exacerbated) temporally associated with the use of IMP. TEAEs are defined as AEs starting after the time of first IMP administration up to and including 8 weeks (56 days) after the final dose.
Time Frame: From Baseline to end of Safety Follow-Up Period (up to Week 31)
Population: Safety set included all randomized study participants who received at least one dose of IMP.
Measure: Number; unit: Percentage of participants
Arm/Group | Placebo | Rozanolixizumab
Number analyzed (Participants) | 10 | 20
Percentage of participants | 0 | 10.0

ADVERSE EVENTS:
Time Frame: From Baseline to end of Safety Follow-Up Period (up to Week 31)
Description: TEAEs are defined as AEs starting after the time of first IMP administration up to and including 8 weeks (56 days) after the final dose. TEAEs were analyzed for Safety Set.
Arm/Group | Placebo | Rozanolixizumab
All-Cause Mortality (participants affected / at risk) | 0/10 | 0/20
Serious Adverse Events (participants affected / at risk) | 1/10 | 5/20
Other Adverse Events (participants affected / at risk) | 6/10 | 18/20
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=10) | Rozanolixizumab (N=20)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1)
Pneumonia viral (Infections and infestations) | 0 (0) | 1 (1)
Head injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Limb injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Skin injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Platelet count decreased (Investigations) | 1 (1) | 1 (1)
Headache (Nervous system disorders) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 0 (0) | 1 (1)
Urticaria (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=10) | Rozanolixizumab (N=20)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 2 (2)
Hypofibrinogenaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Eye pain (Eye disorders) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 3 (3)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 2 (3)
Gingival bleeding (Gastrointestinal disorders) | 0 (0) | 2 (3)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 1 (1)
Constipation (Gastrointestinal disorders) | 1 (1) | 1 (1)
Abdominal distension (Gastrointestinal disorders) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 6 (22)
Fatigue (General disorders) | 0 (0) | 2 (4)
Asthenia (General disorders) | 1 (1) | 1 (4)
Infusion site pain (General disorders) | 1 (1) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 1 (1) | 2 (2)
COVID-19 (Infections and infestations) | 1 (1) | 1 (1)
Urinary tract infection (Infections and infestations) | 1 (1) | 1 (1)
Pharyngitis (Infections and infestations) | 1 (1) | 0 (0)
Platelet count decreased (Investigations) | 1 (1) | 0 (0)
White blood cell count increased (Investigations) | 1 (1) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hyperkalaemia (Metabolism and nutrition disorders) | 1 (4) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (3)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (3)
Headache (Nervous system disorders) | 2 (2) | 12 (25)
Somnolence (Nervous system disorders) | 1 (1) | 0 (0)
Insomnia (Psychiatric disorders) | 1 (1) | 1 (1)
Haematuria (Renal and urinary disorders) | 0 (0) | 2 (2)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Urticaria (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2)
Petechiae (Skin and subcutaneous tissue disorders) | 1 (2) | 1 (2)
Blister (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Hirsutism (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Haemorrhage (Vascular disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (2):
  • Study Protocol (2021-12-06): https://cdn.clinicaltrials.gov/large-docs/88/NCT04224688/Prot_000.pdf
  • Statistical Analysis Plan (2022-08-16): https://cdn.clinicaltrials.gov/large-docs/88/NCT04224688/SAP_001.pdf